CLINICAL TRIAL: NCT01011205
Title: A Multicenter, Three Arm, Randomized, Open Label Clinical Study to Compare Renal Function in Liver Transplant Recipients Receiving an Immunosuppressive Regimen of Advagraf (Immediately or Delayed Post-transplant) and MMF With or Without a Monoclonal Anti-IL2R Antibody (Basiliximab)
Brief Title: Phase 3b Study to Evaluate Advagraf in Combination With Mycophenolate Mofetil and Basiliximab in Liver Transplantation
Acronym: DIAMOND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMR-EC-1106; 2008-002231-32 (EudraCT Number: EudraCT); 2010-021075-89 (EudraCT Number)
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Liver Transplantation
Keywords: Immunosuppression; Liver; Transplant; Advagraf
MeSH Terms: interventions — Mycophenolic Acid; Basiliximab; Adrenal Cortex Hormones; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dosing Regimen 1 (Experimental): Advagraf + MMF + Corticosteroids (Bolus)
  Interventions: Drug: Advagraf; Drug: Mycophenolate Mofetil; Drug: Corticosteroids
- Dosing Regimen 2 (Experimental): Advagraf + MMF + Basiliximab + Corticosteroids (Bolus)
  Interventions: Drug: Advagraf; Drug: Mycophenolate Mofetil; Drug: Basiliximab; Drug: Corticosteroids
- Dosing Regimen 3 (Experimental): Advagraf (5 days delay) + MMF + Basiliximab + Corticosteroids (Bolus)
  Interventions: Drug: Advagraf; Drug: Mycophenolate Mofetil; Drug: Basiliximab; Drug: Corticosteroids

INTERVENTIONS:
Drug: Advagraf — Capsule
  Other Names: MR4; FK506E; tacrolimus modified release
Drug: Mycophenolate Mofetil — Solution for infusion
  Other Names: MMF
Drug: Basiliximab — IV infusion
  Other Names: Simulect
  Arms: Dosing Regimen 2; Dosing Regimen 3
Drug: Corticosteroids — IV bolus
  Other Names: Methylprednisolone or equivalent

SUMMARY:
Comparison of 3 dosing regimens of Advagraf to determine if there is a dosing regimen which may have the potential to cause fewer kidney problems.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing orthotopic liver or split liver allograft transplantation
* Female subject of childbearing potential must have a negative serum or urine pregnancy test at enrollment and must agree to maintain effective birth control during the study

Exclusion Criteria:

* Receiving a multi-organ transplant or having previous received an organ transplant (including liver re-transplantation)
* Receiving an auxiliary graft or in whom a bio-artificial liver (cell system) has been used
* Receiving ABO incompatible graft or a graft from a non heart beating donor
* Ongoing dosing with systemic corticosteroids
* Subjects with systemic infection requiring treatment except viral hepatitis
* Diagnosis of new-onset malignancy prior to transplantation, with the exception of basocellular or squamous cell carcinoma of the skin which had been treated successfully. However, subjects with primary liver carcinoma can be included if they meet the following criteria:

  * < 3 nodes
  * no node larger than 5 cm
  * no metastases
  * no vascular tumoral invasion
* Significant, uncontrolled concomitant infections and/or severe diarrhea, vomiting, active upper gastro-intestinal tract malabsorption or active peptic ulcer
* Subject or donor known to be HIV positive
* Known allergy or intolerance to tacrolimus, macrolide antibiotics, corticosteroids, basiliximab or mycophenolate mofetil or any of the product excipients
* Pregnant woman or breast-feeding mother
* Currently participating in another clinical trial, and/or has taken an investigational drug within 28 days prior to enrollment
* Unlikely to comply with the Visits scheduled in the protocol
* Any unstable medical condition that could interfere with the study objectives in the opinion of the Investigator
* Receiving prohibited concomitant therapy, or received prohibited concomitant therapy within 28 days prior to enrollment
* Any form of substance abuse, psychiatric disorder or condition which, in the opinion of the Investigator, may complicate communication with the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 893 (Actual)
Dates: Start 2009-09-30 (Actual); Primary Completion 2013-01-04 (Actual); Study Completion 2013-01-04 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration rate (GFR) at 24 Weeks after transplantation estimated using the MDRD4 formula | 24 weeks

SECONDARY OUTCOMES:
Incidence of and time to first incidence of the composite event: graft loss (defined as re-transplantation or death) or biopsy confirmed acute rejection (BCAR) | 24 weeks
GFR at 24 Weeks after transplantation measured by Iothalamate clearance | 24 weeks
GFR at 24 Weeks after transplantation estimated using a Cystatin C based formula | 24 weeks
Creatinine clearance at 24 Weeks after transplantation estimated using the Cockcroft and Gault formula | 24 weeks
Incidence of and time to first incidence of acute rejection | 24 weeks
Incidence of and time to first incidence of corticosteroid-resistant acute rejection | 24 weeks
Overall frequency of acute rejection episodes | 24 weeks
Incidence of and time to first incidence of biopsy confirmed acute rejection | 24 weeks
Incidence of and time to first incidence of biopsy confirmed corticosteroid-resistant acute rejection | 24 weeks
Overall frequency of biopsy confirmed acute rejection episodes | 24 weeks
Severity of biopsy confirmed acute rejection episodes | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Global Development - EU
Locations (72):
- 160, Buenos Aires, Argentina
- 001, Innsbruck, Austria
- 146, Minsk, Belarus
- Belgium (4):
  - 008, Brussels
  - 006, Ghent
  - 009, Leuven
  - 010, Liège
- 163, São Paulo, Brazil
- Canada (5):
  - 153, Edmonton
  - 150, Halifax
  - 151, London
  - 152, Montreal
  - 154, Vancouver
- 169, Bogata, Colombia
- 147, Prague, Czechia
- 026, Helsinki, Finland
- France (14):
  - 041, Besançon
  - 157, Bordeaux
  - 043, Caen
  - 031, Créteil
  - 039, Lyon
  - 045, Marseille
  - 158, Montpelier
  - 037, Nice
  - 042, Paris
  - 044, Paris
  - 035, Paris
  - 038, Strasbourg
  - 033, Toulouse
  - 034, Villejuif
- Germany (12):
  - 056, Berlin
  - 058, Erlangen
  - 051, Frankfurt
  - 055, Göttingen
  - 057, Hanover
  - 142, Jena
  - 053, Kiel
  - 054, Leipzig
  - Site: 156, Mainz
  - 052, Münster
  - 060, Regensberg
  - 059, Tübingen
- 061, Budapest, Hungary
- 070, Dublin, Ireland
- Italy (8):
  - 073, Bergamo
  - 075, Bologna
  - 076, Genova
  - 077, Naples
  - 079, Naples
  - 072, Padua
  - 074, Rome
  - 071, Udine
- Site: 166, Mexico City, Mexico
- Poland (2):
  - 086, Warsaw
  - 087, Warsaw
- 091, Bucharest, Romania
- Russia (2):
  - 096, Moscow
  - 097, Moscow
- 148, Johannesburg, South Africa
- Spain (8):
  - 114, A Coruña
  - 109, Barcelona
  - 106, Barcelona
  - 110, Barcelona
  - 115, Madrid
  - 108, Madrid
  - 117, Madrid
  - 116, Zaragoza
- 126, Gothenberg, Sweden
- 131, Zurich, Switzerland
- United Kingdom (3):
  - 136, Birmingham
  - 171, Leeds
  - 138, London

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=57